CLINICAL TRIAL: NCT03270358
Title: OStéopontin as a Marker Of StenoSIS - OSMOSIS
Acronym: OSMOSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-AOI-03
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Stenosis
MeSH Terms: conditions — Constriction, Pathologic | interventions — Blood Specimen Collection; Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with stenosis (Experimental): Patient coming to the vascular surgery unit to receive surgery regarding their fistula stenosis
  Interventions: Procedure: Blood sampling in arterioveinous fistula with stenosis
- patient without stenosis (Other): Patient coming for their dialysis
  Interventions: Procedure: Blood sampling in arterioveinous fistula without stenosis

INTERVENTIONS:
Procedure: Blood sampling in arterioveinous fistula without stenosis — Plasmatic osteopontin level (ng/ml) collected in the patient's arteriovenous fistula.
  Blood sampling in arterioveinous fistula right before a dialysis session
  Arms: patient without stenosis
Procedure: Blood sampling in arterioveinous fistula with stenosis — Blood sampling in arterioveinous fistula right before the surgery for stenosis of the fistula
  Arms: patient with stenosis

SUMMARY:
Our hypothesis is that a plasma protein named osteopontin (OPN) could serve as a biological predictive marker of acute AVF dysfunction. In several scientific studies, plasma OPN was correlated with coronary stent restenosis, and with cardiovascular outcome in patients with diabetes and renal insufficiency. This protein is secreted by several cellular types, like distal tubule epithelial cells, macrophages, but also fibroblasts and cardiac and vascular endothelial cells, in response to several specific stimuli. It acts like a cytokine, inducing immunological mechanisms as well as tissue remodeling.

The main objective of this study is to show that the amount of plasma OPN is higher in patients presenting with an AVF stenosis, compared with patients with a functioning AVF.

OSMOSIS is a monocentric pilot study that will include patients into two groups during 12 months (no specific follow-up). The control group will include patients that have been dialyzed on an AVF, in the dialysis center of Nice University Hospital, for at least 3 months without any incident. The experimental group will include hemodialysis patients hospitalized in the department of vascular surgery for acute AVF dysfunction, needing endovascular or open surgical revision for venous stenosis.

Blood will be withdrawn right before dialysis or surgical procedure. Plasma OPN will me measured by ELISA. Their clinical data would be collected from medical file at the same time. After the procedure, patients will be followed-up according to usual protocols.

To show a significant difference of 100ng/mL plasma OPN between the two groups, with a power of 90% and alpha risk of 0.05, we plan to include 76 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients under a social security scheme
* Written informed consent obtain
* 18 years old or older
* end-stage renal failure disease with 3 months dialysis minimum on a native arteriovenous fistula

Non-inclusion Criteria:

* Subject under juridicial protection
* Pregnant or lactating women
* Subject already enrolled in a clinical trial involving a drug or an implantable medical device

Exclusion Criteria:

* Withdrawal of consent
* Investigator or sponsor decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Plasmatic osteopontin level | at inclusion
  Plasmatic osteopontin level (ng/ml) collected in the patient's arteriovenous fistula.
  * Control arm: right before a dialysis session
  * Experimental arm: right before the surgery for stenosis of the fistula

SECONDARY OUTCOMES:
Peripheral plasmatic osteopontin level in the contralateral arm | at inclusion
  Peripheral plasmatic osteopontin level (ng/ml) collected in the contralateral arm (to measure the potential bias of a local osteopontin production in the fistula)
Peripheral plasmatic osteopontin level in the contralateral arm | at inclusion
  Measure of the plasmatic osteopontin specificity and sensibility on the occurrence of a fistula stenosis (differents tresholds)
Peripheral plasmatic osteopontin level in the contralateral arm | at inclusion
  Collection of comorbidity factors (diabetes, arterial hypertension, coronaropathy, overweight (BMI)), clinical factors (age and gender) and treatments at the time of patient's inclusion (anticoagulant, antisludge, antihypertensive drug, statins, erythropoietin)

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana SADAGHIANLOO, Principal Investigator — sadaghianloo.n@chu-nice.fr
Locations (1):
- CHU de Nice - Service de chirurgie vasculaire, Nice, France